CLINICAL TRIAL: NCT01135992
Title: A Trial Assessing the Implications of Switching From Insulin Glargine to Insulin Degludec in Subjects With Type 2 Diabetes Mellitus (BEGIN™: SIMPLIFY)
Brief Title: Switching From Insulin Glargine to Insulin Degludec in Subjects With Type 2 Diabetes Mellitus (BEGIN™)
Acronym: BEGIN™
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NN1250-3839; U1111-1114-8802 (Other: WHO)
Record Dates: First submitted 2010-05-31; First posted 2010-06-03 (Estimated); Results first posted 2016-01-22 (Estimated); Last update posted 2016-01-22 (Estimated); Status verified 2015-12

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin degludec; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IGlar/IDeg (Experimental)
  Interventions: Drug: insulin glargine
- IDeg 3TW (Experimental)
  Interventions: Drug: insulin degludec

INTERVENTIONS:
Drug: insulin degludec — Individually adjusted insulin degludec administered three times weekly with continued unchanged pre-trial OAD (oral anti-diabetic drug) treatment for 12 weeks
  Arms: IDeg 3TW
Drug: insulin glargine — Subjects continue their pre-trial insulin glargine once daily plus OAD (oral anti-diabetic drug) treatment for four weeks before switch to insulin degludec
  Arms: IGlar/IDeg

SUMMARY:
This trial is conducted in the United States of America (USA). The aim of this clinical trial is to assess the implications of switching from insulin glargine (IGlar) to insulin degludec (IDeg) in subjects with type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus (diagnosed clinically) for at least 6 months
* HbA1c maximum 10 % by central laboratory analysis
* Current treatment with basal-oral therapy (BOT) (no prandial insulin ever) consisting of: at least three months with insulin glargine once daily (average prescribed dose must have been unchanged (within plus/minus 10%) for four weeks prior to Visit 1 as confirmed by patient records or verbal confirmation by the subject) in combination with stable (unchanged doses for at least 3 months prior to Visit 1) OAD (metformin, insulin secretagogues, pioglitazone, sitagliptin or alpha-glucosidase-inhibitor) treatment in any approved (according to label) dose or combination

Exclusion Criteria:

* Use within the last three months prior to Visit 1 of: Exenatide, Liraglutide or Thiazoledinediones (TZDs) other than Pioglitazone
* Cardiovascular disease (CVD) defined as: stroke; decompensated heart failure New York Heart Association (NYHA) class III or IV; myocardial infarction; unstable angina pectoris; or coronary arterial bypass graft or angioplasty within the last six months prior to Visit 1
* Recurrent severe hypoglycaemia (more than one severe hypoglycaemic episode during the last 12 months), or hypoglycaemic unawareness as judged by the Investigator, or hospitalisation for diabetic ketoacidosis during the previous six months
* Pregnancy, breast-feeding, the intention of becoming pregnant or not using adequate contraceptive measures according to local requirements
* Previous participation in this trial. Participation is defined as started on trial medication. Rescreening of screening failures is allowed only once within the limits of the recruitment period
* Known or suspected hypersensitivity to trial products or related products

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2010-06; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (26):
- United States (26):
  - Novo Nordisk Clinical Trial Call Center, Goodyear, Arizona
  - Novo Nordisk Clinical Trial Call Center, Phoenix, Arizona
  - Novo Nordisk Clinical Trial Call Center, Anaheim, California
  - Novo Nordisk Clinical Trial Call Center, Chino, California
  - Novo Nordisk Clinical Trial Call Center, Concord, California
  - Novo Nordisk Clinical Trial Call Center, Fresno, California
  - Novo Nordisk Clinical Trial Call Center, Greenbrae, California
  - Novo Nordisk Clinical Trial Call Center, Palm Springs, California
  - Novo Nordisk Clinical Trial Call Center, Kissimmee, Florida
  - Novo Nordisk Clinical Trial Call Center, Chicago, Illinois
  - Novo Nordisk Clinical Trial Call Center, Metairie, Louisiana
  - Novo Nordisk Clinical Trial Call Center, Omaha, Nebraska
  - Novo Nordisk Clinical Trial Call Center, Henderson, Nevada
  - Novo Nordisk Clinical Trial Call Center, Dover, New Hampshire
  - Novo Nordisk Clinical Trial Call Center, Nashua, New Hampshire
  - Novo Nordisk Clinical Trial Call Center, Lawrenceville, New Jersey
  - Novo Nordisk Clinical Trial Call Center, Toms River, New Jersey
  - Novo Nordisk Clinical Trial Call Center, Albany, New York
  - Novo Nordisk Clinical Trial Call Center, Charlotte, North Carolina
  - Novo Nordisk Clinical Trial Call Center, Melrose Park, Pennsylvania
  - Novo Nordisk Clinical Trial Call Center, Pittsburgh, Pennsylvania
  - Novo Nordisk Clinical Trial Call Center, Chattanooga, Tennessee
  - Novo Nordisk Clinical Trial Call Center, Kingsport, Tennessee
  - Novo Nordisk Clinical Trial Call Center, Austin, Texas
  - Novo Nordisk Clinical Trial Call Center, Fort Worth, Texas
  - Novo Nordisk Clinical Trial Call Center, Olympia, Washington

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 27 sites in the United States of America (U.S.)
Pre-assignment Details: The trial was conducted on subjects with type 2 diabetes mellitus currently treated with IGlar once daily (OD) and oral antidiabetic drug (OAD) therapy.
Groups:
- IGlar/IDeg: Subjects received 4 weeks of unchanged pre-trial insulin glargine (IGlar) once daily (OD) followed by 12 weeks of insulin degludec (IDeg) 200 U/mL 3 times weekly (3TW) subcutaneously, both in combination with unchanged pre-trial oral antidiabetic drug [OAD] treatment.
Period: Overall Study
Arm/Group | IGlar/IDeg
Started | 143
Exposed | 142 (One subject was withdrawn before being exposed.)
Full Analysis Set | 129
Completed | 122
Not Completed | 21
Not completed — Adverse Event | 1
Not completed — Lack of Efficacy | 1
Not completed — Protocol Violation | 2
Not completed — Withdrawal criteria | 10
Not completed — Unclassified | 7

BASELINE CHARACTERISTICS:
Population: Full Analysis set (FAS)-Includes 129 subjects only as 13 subjects did not receive IDeg.
Arm/Group | IGlar/IDeg
Number analyzed (Participants) | 129
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.7 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43
  Male | 86
HbA1c (glycosylated haemoglobin) at baseline [Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin] | 7.5 (1.1)
Fasting plasma glucose (FPG) at baseline [Mean (Standard Deviation); unit: mmol/L] | 7.0 (2.2)
Body weight at baseline [Mean (Standard Deviation); unit: kg] | 99.3 (20.4)

OUTCOME MEASURES:

1. Primary Outcome: HbA1c (Glycosylated Haemoglobin)
Description: HbA1C at week 4 and 16
Time Frame: Week 4 and Week 16
Population: FAS (Full Analysis Set) includes all subjects that were switched to IDeg 3TW treatment
Measure: Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin
Arm/Group | IGlar/IDeg
Number analyzed (Participants) | 129
percentage of glycosylated haemoglobin
  Week 4 (N=128) (IGlar) | 7.4 (1.0)
  Week 16 (N=122)(IDeg) | 7.2 (1.1)

2. Secondary Outcome: Fasting Plasma Glucose (FPG)
Description: FPG at week 4 and 16
Time Frame: Week 4 and Week 16
Population: FAS (Full Analysis Set) includes all subjects that were switched to IDeg 3TW treatment
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | IGlar/IDeg
Number analyzed (Participants) | 129
mmol/L
  Week 4 (N=128) (IGlar) | 7.0 (2.3)
  Week 16 (N=122) (IDeg) | 6.3 (2.2)

3. Secondary Outcome: Change in Body Weight
Description: Change from baseline in body weight after week 4 and after week 16
Time Frame: Week 0, Week 4, Week 16
Population: Safety Analysis Set includes all subjects who received at least one dose of the investigational product or its comparator. Missing data is imputed using LOCF (last observation carried forward)
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | IGlar/IDeg
Number analyzed (Participants) | 142
kg
  Week 4(N= 142) (IGlar) | 0.1 (0.4)
  Week 16 (N=129) (IDeg) | 0.6 (2.2)

4. Secondary Outcome: Rate of Treatment Emergent Adverse Events (AEs)
Description: Corresponds to rate of AEs per 100 patient years of exposure. Mild AEs: no or transient symptoms, no interference with subject's daily activities. Moderate AEs: marked symptoms, moderate interference with subject's daily activities. Severe AEs: considerable interference with subject's daily activities, unacceptable. Serious adverse event (SAE): AE that at any dose results in any of the following: death, a life-threatening experience, in-subject hospitalization/prolongation of existing hospitalisation, persistent/significant disability/incapacity/congenital anomaly/birth defect
Time Frame: Weeks 0-4 (IGlar), Weeks 4-16 (IDeg 3TW)
Population: Safety Analysis Set includes all subjects who received at least one dose of the investigational product or its comparator.
Measure: Number; unit: events per 100 patient years
Arm/Group | IGlar/IDeg
Number analyzed (Participants) | 142
events per 100 patient years
  Adverse events (N=142)(week 4)(IGlar) | 370
  Serious AEs (N=142 ) (week 4)(IGlar) | 9
  Severe AEs (N=142)(week 4) (IGlar) | 19
  Moderate AEs (N=142) (week 4)(IGlar) | 102
  Mild AEs (N=142)(week 4) (IGlar) | 250
  Fatal AEs (N=142) (week 4) (IGlar) | 0
  Adverse events (N=129) (week 16) (IDeg) | 424
  Serious AEs (n=129) (week 16) (IDeg) | 7
  Severe AEs (N=129) (week 16) (IDeg) | 10
  Moderate AEs (N=129) (week 16) (IDeg) | 132
  Mild AEs (N=129) (week 16) (IDeg) | 280
  Fatal AEs (N=129) (week 16) (IDeg) | 0
  Adverse Events (N=142) (Total) | 409
  Serious AEs (N=142) (Total) | 8
  Severe AEs (N=142) (Total) | 13
  Moderate AEs (N=142) (Total) | 124
  Mild AEs (N=142) (Total) | 273
  Fatal AEs (N=142)(Total) | 0

5. Secondary Outcome: Rate of Confirmed Hypoglycaemic Episodes
Description: Rate of confirmed hypoglycaemic episodes per 100 patient years of exposure (PYE). Confirmed hypoglycaemic episodes consisted of severe hypoglycaemia as well as minor hypoglycaemic episodes with a confirmed plasma glucose value of less than 3.1 mmol/L.
Time Frame: Weeks 0-4 (IGlar), Weeks 4-16 (IDeg 3TW)
Population: as for outcome 4
Measure: Number; unit: episodes per 100 patient years
Arm/Group | IGlar/IDeg
Number analyzed (Participants) | 142
episodes per 100 patient years
  IGlar (N=142) (week 4) | 453
  IDeg (N=129) (week 16) | 424

6. Secondary Outcome: Rate of Nocturnal Confirmed Hypoglycaemic Episodes
Description: Rate of nocturnal confirmed hypoglycaemic episodes per 100 patient years of exposure (PYE). Confirmed hypoglycaemic episodes consisted of severe hypoglycaemia as well as minor hypoglycaemic episodes with a confirmed plasma glucose value of less than 3.1 mmol/L. Nocturnal hypoglycaemic episodes are defined as occuring between 00:01 and 05:59 a.m.
Time Frame: Weeks 0-4 (IGlar), Weeks 4-16 (IDeg 3TW)
Population: as for outcome 4
Measure: Number; unit: episodes per 100 patient years
Arm/Group | IGlar/IDeg
Number analyzed (Participants) | 142
episodes per 100 patient years
  IGlar (week 4) (N=142) | 111
  IDeg (week 16) (N=129) | 83

ADVERSE EVENTS:
Time Frame: The adverse events were collected in a time frame of 0-4 weeks (IGlar) and 4-16 weeks (IDeg 3TW)
Description: Safety analysis set includes all subjects who received at least one dose of the investigational product or its comparator
Arm/Group | IGlar/IDeg
Serious Adverse Events (participants affected / at risk) | 3/142
Other Adverse Events (participants affected / at risk) | 0/142
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | IGlar/IDeg (N=142)
Cholelithiasis (IGlar) (Hepatobiliary disorders) | 0 (0) — (week 4) (N=142)
Cholelithiaisis (IDeg) (Hepatobiliary disorders) | 1/129 (1) — (week 16) (N=129)
Cholelithiasis (Total) (Hepatobiliary disorders) | 1 (1) — (N=142)
Lumbar spinal stenosis (IGlar) (Musculoskeletal and connective tissue disorders) | 1 (1) — (week 4) (N=142)
Lumbar spinal stenosis (IDeg) (Musculoskeletal and connective tissue disorders) | 0/129 (0) — (week 16) (N=129)
Lumbar spinal stenosis (Total) (Musculoskeletal and connective tissue disorders) | 1 (1) — (N=142)
Carotid artery occlusion (IGlar) (Nervous system disorders) | 0 (0) — (week 4)(N=142)
Carotid artery occlusion (IDeg) (Nervous system disorders) | 1/129 (1) — (week 16)(N=129)
Carotid artery occlusion (Total) (Nervous system disorders) | 1 (1) — (N=142)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk maintains the right to be informed of any Investigator plans for publication and to review any scientific paper, presentation, communication or other information concerning the investigation described in this protocol. Any such communication must be submitted in writing to the Novo Nordisk trial manager prior to submission for comments. Comments will be given within four weeks from receipt of the planned communication.